CLINICAL TRIAL: NCT03399435
Title: An Exploratory Phase I Randomized, Single-site, Double-blind, Active-controlled, Parallel-group, Single-administration, Dose-escalation Trial to Investigate the Safety and Tolerability of Neosaxitoxin Alone and in Combination With Bupivacaine (With and Without Epinephrine), in Perineural Administrations for Brachial Plexus Blockade in Healthy Subjects
Brief Title: A Study in Healthy Male Volunteers to Investigate the Safety and Tolerability of a Single Dose of Neosaxitoxin Alone and in Combination With Bupivacaine (With and Without Epinephrine) for Brachial Plexus Blockade
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor decided to stop further dosing of healthy volunteers after reviewing the obtained efficacy data. The decision is not related to any safety concern.
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HP7020-02; 2016-003958-33 (EudraCT Number); U1111-1189-1950 (Registry Identifier: World Health Organization)
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Anesthesia; Anesthesia, Local; Analgesia
Keywords: Regional anesthesia; Brachial plexus blockade; Sensory and motor function testing
MeSH Terms: conditions — Agnosia | interventions — Epinephrine; neosaxitoxin; Triiodothyronine

STUDY DESIGN:
Intervention Model Description: Part A: 8 cohorts (equivalent to 40 subjects) are planned to be treated with ascending doses of neosaxitoxin combined with fixed doses of bupivacaine and epinephrine.
  Part B: Part B will start at the earliest after 4 cohorts of Part A have been treated. Ascending doses of neosaxitoxin combined with fixed doses of bupivacaine.
  Part C: Part C will comprise 4 treatment groups in which all participants will receive the same neosaxitoxin dose alone, or neosaxitoxin combined with epinephrine, or neosaxitoxin combined with bupivacaine with or without epinephrine.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sponsor, personnel of the central research pharmacy at the site, the pharmacy CRA and the bioanalytical lab are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental): 8 cohorts are planned to be treated.
  Interventions: Combination Product: Neosaxitoxin combined with bupivacaine low and epinephrine (T1); Combination Product: Bupivacaine low combined with epinephrine (C1); Combination Product: Bupivacaine high combined with epinephrine (C2)
- Part B (Experimental): Part B will start at the earliest after 4 cohorts of Part A have been treated. Up to 8 cohorts are planned to be treated.
  Interventions: Combination Product: Neosaxitoxin combined with bupivacaine low (T2); Drug: Bupivacaine low (C3); Drug: Bupivacaine high (C4)
- Part C (Experimental): Part C will comprise 4 treatment groups. The neosaxitoxin dose will be the same in all 4 treatment groups.
  Interventions: Drug: Neosaxitoxin (T3); Combination Product: Neosaxitoxin combined with epinephrine (T4); Combination Product: Neosaxitoxin combined with bupivacaine low and epinephrine; Combination Product: Neosaxitoxin combined with bupivacaine low

INTERVENTIONS:
Combination Product: Neosaxitoxin combined with bupivacaine low and epinephrine (T1) — A single injection: Neosaxitoxin from 1.25 to 60 µg. Bupivacaine 40 mg. Epinephrine 100 µg.
  Arms: Part A
Combination Product: Bupivacaine low combined with epinephrine (C1) — A single injection: Bupivacaine 40 mg. Epinephrine dose 100 µg.
  Arms: Part A
Combination Product: Bupivacaine high combined with epinephrine (C2) — A single injection: Bupivacaine 100 mg. Epinephrine 100 µg.
  Arms: Part A
Combination Product: Neosaxitoxin combined with bupivacaine low (T2) — A single injection: Neosaxitoxin from 1.25 to 60 μg. Bupivacaine from 10 to 80 mg.
  Arms: Part B
Drug: Bupivacaine low (C3) — A single injection: Bupivacaine from 10 to 80 mg.
  Arms: Part B
Drug: Bupivacaine high (C4) — A single injection: Bupivacaine 100 mg.
  Arms: Part B
Drug: Neosaxitoxin (T3) — A single injection: Neosaxitoxin will be between 1.25 and 60 µg.
  Arms: Part C
Combination Product: Neosaxitoxin combined with epinephrine (T4) — A single injection: Neosaxitoxin will be between 1.25 and 60 μg. Epinephrine 100 µg.
  Arms: Part C
Combination Product: Neosaxitoxin combined with bupivacaine low and epinephrine — A single injection: Neosaxitoxin will be between 1.25 to 60 µg. Bupivacaine dose based on results from Part B (10 to 80 mg). Epinephrine 100 µg.
  Arms: Part C
Combination Product: Neosaxitoxin combined with bupivacaine low — A single injection: Neosaxitoxin will be between 1.25 to 60 μg. Bupivacaine dose based on results from Part B (10 to 80 mg).
  Arms: Part C

SUMMARY:
Neosaxitoxin is a new compound that is in clinical development as local anesthetic for surgical anesthesia and postoperative analgesia.

The primary objective of this study is to evaluate the systemic and local safety and tolerability of ascending doses of neosaxitoxin alone and in combination with fixed doses of bupivacaine (with and without epinephrine), following brachial plexus blockade in healthy male subjects.

Secondary objectives:

* Evaluate the pharmacodynamics (PD) of ascending doses of neosaxitoxin, alone and in combination with fixed doses of bupivacaine (with and without epinephrine), following brachial plexus blockade.
* Characterize the pharmacokinetics (PK) of neosaxitoxin and bupivacaine after brachial plexus blockade with neosaxitoxin alone or different drug combinations: neosaxitoxin and epinephrine, neosaxitoxin and bupivacaine, or neosaxitoxin and bupivacaine and epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent to participate.
* Male subject, aged 18 years to 55 years, inclusive.
* Body mass index between 20.0 kg/m2 and 30.0 kg/m2 inclusive, with a minimal body weight of 60.0 kg.
* Subject must be in good health as determined by the prior/concomitant diseases, physical and laboratory examinations.
* Subject must be willing not to donate sperm and to use barrier contraception (condom) during sexual intercourse with women from the administration of IMP until Day 90 since IMP administration. The subject must be willing to ensure that the female sexual partner of childbearing potential uses at least 1 additional method of contraception with a low failure rate defined as <1% per year (e.g., oral contraceptives) during this time frame. A single barrier method alone is not acceptable.

Exclusion Criteria:

At enrollment:

* Resting pulse rate <50 beats or >90 beats per minute.
* Resting systolic blood pressure <90 mmHg or >140 mmHg. Resting diastolic blood pressure >90 mmHg.
* Prolongation of QTcF at enrollment, i.e., QTcF >450 ms, or presence of any other of risk factors for torsade de pointes or other disturbances of cardiac de- and repolarization.
* Any out-of-reference range value for the following safety laboratory parameters: GGT, serum creatinine, PT, and INR.
* Any exclusion range met for urinalysis and the following safety laboratory parameters: ALT, AST, ALP, total bilirubin, glucose, LDH, potassium, total protein, sodium, calcium, CK, hemoglobin, hematocrit, white blood cell count, and platelets.
* Any out-of-reference range value for any other safety laboratory parameter that is judged as clinically relevant by the investigator.
* Positive or missing virus serology test for HIV Type 1 or Type 2 antibodies and antigen, hepatitis B surface antigen, hepatitis B core antibodies, or hepatitis C virus antibodies.
* Subject received IMP in another clinical trial within 1 month before the Enrollment Visit. Depending on the nature of the previous IMP, a longer washout may be needed.
* Diseases or conditions known to interfere with the distribution, metabolism, or excretion of drugs.
* History of orthostatic hypotension.
* History of, or at risk of seizures.
* Significant cardiovascular, respiratory, neuromuscular diseases, or other systemic illness.
* Subject with an oxygen saturation of less than 95%, as measured by pulse oximetry, or subject with known or suspected respiratory difficulty or any condition that may compromise a subject's breathing or ability to maintain adequate oxygen saturation.
* Known vocal chord palsy.
* Any relevant symptom of neurological dysfunction of the motor and sensory system based on sensory and motor function testing. History or presence of symptoms of depression or anxiety disorders.
* Previous injury or surgery of the involved shoulder in the last 2 years.
* Any relevant local abnormality at the targeted area of injection.
* Any acute or chronic pain condition requiring ongoing treatment or limiting daily activities.
* Definite or suspected history of drug allergy, particularly to bupivacaine or other local anesthetics, epinephrine, or clinically relevant other allergies.
* Evidence or history of alcohol or drug abuse including positive or missing drugs of abuse screen.
* Regular use of any medication, including herbal remedies or over-the counter medication within 2 weeks before enrollment into this trial and anticipated use during the course of the trial.
* Habitually smoking more than 10 cigarettes, 2 cigars, or 2 pipes of tobacco per day within the last 6 months before enrollment in this trial.
* Known or suspected of not being able to comply with the requirements of the trial protocol or the instructions of the trial site staff.
* Not able to communicate meaningfully with the trial site staff.
* Employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site, as well as family members of the employees or the investigator.
* Blood loss of 500 mL or more within 3 months before enrollment in this trial.

On Day -1:

* Any relevant deterioration in the health of the subject since the Enrollment Visit possibly impacting participation in the trial, including AEs, safety laboratory parameters, vital signs, body temperature, ECG, or other safety parameters at the discretion of the investigator.
* Out-of-reference blood pressure or pulse rate if technical failure can be excluded and result is confirmed by at least 1 additional measurement: Systolic blood pressure <90 mmHg or >140 mmHg, diastolic blood pressure >90 mmHg, pulse rate <50 beats or >90 beats per minute.
* Clinically relevant QTcF interval prolongation, i.e., QTcF interval >450 ms.
* Any out-of-reference range value for the following safety laboratory parameters: GGT, serum creatinine, PT, and INR.
* Any exclusion range met for urinalysis and the following safety laboratory parameters: ALT, AST, ALP, total bilirubin, glucose, LDH, potassium, total protein, sodium, calcium, CK, hemoglobin, hematocrit, white blood cell count, and platelets.
* Any out-of-reference range value for any other safety laboratory parameter that is judged as clinically relevant by the investigator.
* Positive or missing drugs of abuse screen.
* Intake of forbidden medication since the enrollment in this trial.
* Participation in another clinical trial since the Enrollment Visit.
* Blood loss of 100 mL or more since enrollment in this trial.
* Failure to comply with trial requirements, e.g., consumption of alcohol, etc., considered by the investigator to affect subject safety or interfere with the integrity of the trial.
* Any relevant local abnormality at the targeted area of injection.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting events (DLEs) in all parts of the trial. | up to 15 days after IMP (investigational medicinal product, i.e. study drug administration)
Occurrence of other adverse events (AEs) leading to premature termination of dose escalation in Part A and Part B. | up to 15 days after IMP administration

SECONDARY OUTCOMES:
Cold detection threshold (CDT). | Baseline, 24 and 48 hours after IMP administration
Warm detection threshold (WDT) | Baseline, 24 and 48 hours after IMP administration
Mechanical detection threshold (MDT) | Baseline, 24 and 48 hours after IMP administration
Cold pain threshold (CPT) | Baseline, 24 and 48 hours after IMP administration
Heat pain threshold (HPT) | Baseline, 24 and 48 hours after IMP administration
Mechanical pain threshold (MPT) | Baseline, 24 and 48 hours after IMP administration
Muscle grip strength (ipsilateral) | Baseline, 24 and 48 hours after IMP administration
Muscle motor function (flexion and extension elbow joint, abduction shoulder joint) | Baseline, 24 and 48 hours after IMP administration
AUC0-t of neosaxitoxin | up to 56 hours after IMP administration
AUC0-t of bupivacaine | up to 56 hours after IMP administration
Cmax of neosaxitoxin | up to 56 hours after IMP administration
Cmax of bupivacaine | up to 56 hours after IMP administration
tmax of neosaxitoxin | up to 56 hours after IMP administration
tmax of bupivacaine | up to 56 hours after IMP administration

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grünenthal GmbH
Locations (1):
- NL001, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site ( according to the EFPIA Data Sharing Principles.
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials